CLINICAL TRIAL: NCT03953742
Title: A Phase 1, First-in-Human Study Evaluating the Safety, Tolerability, and Pharmacokinetics of CPI-200 Via Intravenous Infusion in Patients With Advanced Solid Tumors
Brief Title: Study of CPI-200 in Patients With Advanced Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coordination Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPI-200CL01
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Advanced Solid Tumor
Keywords: Intravenous infusion; Phase 1; CPI-200

STUDY DESIGN:
Intervention Model Description: Accelerated titration method followed by a conventional 3 + 3 study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPI-200 (Experimental): Dose Escalation Group: CPI-200 will be administered via intravenous infusion once every 3 weeks for up to 7 dose levels using an accelerated titration method followed by a conventional 3 + 3 study design
  Dose Expansion Group: Maximum tolerated dose or the recommended Phase 2 dose (RP2D) from dose escalation group
  Interventions: Drug: CPI-200

INTERVENTIONS:
Drug: CPI-200 — CPI-200 will be administered via intravenous infusion on Day 1 of a 21-Day cycle

SUMMARY:
This is a prospective, open-label, single arm, non-randomized study of CPI-200 in patients with advanced tumors. CPI-200 is administered via intravenous infusion using an accelerated titration method followed by a conventional 3 + 3 study design to identify the maximum tolerated dose (MTD)

DETAILED DESCRIPTION:
Primary Objectives:

• To determine the safety, tolerability and maximum tolerated dose (MTD) of CPI-200 in patients with advanced tumors

Secondary Objectives:

* To evaluate the pharmacokinetics (PK) of CPI-200
* To evaluate clinical response and resolution of symptoms after CPI-200 treatment
* To characterize adverse events of CPI-200 in patients with advanced cancers

Up to 7 dose levels of CPI-200 will be tested using an accelerated titration method followed by a conventional 3 + 3 dose escalation study design. MTD will be defined as the dose associated with a dose limiting toxicity (DLT) in less than or equal to 33% of patients at the dose level tested. Dose limiting toxicity (DLT) is defined as one of the following events occurring from the intravenous injection of CPI-200 within 21 days:

* All Grade 4 or greater adverse events as determined by CTCAEv5 criteria, excluding toxicities clearly related to disease progression or inter-current illness
* Any Grade 3 or greater non-hematologic, non-dermatologic toxicity with the exception of Grade 3 nausea, vomiting or diarrhea if lasting less than 72 hours, alopecia, or Grade 3 fatigue if lasting less than 7 days as determined by CTCAEv5 criteria
* Grade 3 thrombocytopenia in the presence of bleeding
* Grade 3 or greater febrile neutropenia
* Any hematologic or non-hematologic adverse events or abnormal laboratory value(s) related to CPI-200 that result(s) in permanent study discontinuation of study treatment

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Males and females
* Have a histologically or cytologically confirmed diagnosis of advanced solid tumor
* Have advanced or metastatic disease refractory to standard curative or palliative therapy or contraindication to standard therapy
* Have an ECOG performance status of 0-1
* Have a life expectancy of at least 12 weeks (in the opinion of the investigator)
* Have adequate bone marrow reserve, liver and renal function
* Be reasonably recovered from preceding major surgery and no major surgery within 4 weeks prior to the start of Day 1 treatment
* Have a negative pregnancy test for females with child bearing age at screening and should not be breast feeding
* Be willing to abstain from sexual activity or practice physical barrier contraception from study entry to 3 months after the last day of treatment

Exclusion Criteria:

* Have peripheral sensory neuropathy of Grade 2 or greater at screening
* Have known hypersensitivity to chemotherapeutic agents
* Have thrombocytopenia with complications including hemorrhage or bleeding > Grade 2 that required medical intervention or any hemolytic condition or coagulation disorders that would make participation unsafe
* Have unresolved toxicity from previous treatment or previous investigational agents; excluding alopecia
* Received investigational agents or systemic anticancer agents (other than neurotoxic compounds) within 5 half lives or 28 days, whichever is shorter, prior to Day 1 of treatment
* Have signs or symptoms of end organ failure, major chronic illnesses other than cancer, or any severe concomitant conditions
* Have experienced any of the following within the 6-month period prior to screening: unstable angina, myocardial infarction or cerebrovascular accident, transient ischemic attack, cardiac failure with known ejection fraction less than 40%
* Have other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that would make the patient inappropriate for enrollment in this study
* Is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 21 days
  • To determine the maximum tolerated dose (MTD), which is defined as the dose level at which fewer than 33% of patients experience a dose limiting toxicity (DLT) using a 3+3 strategy as assessed by CTCAE

SECONDARY OUTCOMES:
Rate of Clinical Benefit | through study completion, an average of 4 months
  • To assess clinical benefit by response rate and resolution of symptoms, which will be reported as response rate (%) of participants
Rate of Adverse Effect | through study completion, an average of 4 months
  • To assess adverse effect as either treatment-related or non-treatment-related as defined by CTCAE, which will be reported as % of participants
Maximum Plasma Concentration (Cmax) | 8 Days
  • To evaluate maximum plasma concentration (Cmax) of CPI-200 in patients tested
Area Under the Curve (AUC) | 8 Days
  • To evaluate area under the curve (AUC) of CPI-200 in patients tested

CONTACTS AND LOCATIONS:
Locations (1):
- South Texas Accelerated Research Therapeutics (START Midwest), Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
The data will not be shared due to confidentiality agreements.